CLINICAL TRIAL: NCT07086521
Title: A Phase 1, Double-blinded, Randomized, Dose-repeating, Placebo-controlled, Cross-over Study to Assess the Safety and Preliminary Efficacy of Allogeneic ULSC on Disease Severity in Facioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: Safety and Preliminary Efficacy of ULSC in Facioscapulohumeral Muscular Dystrophy (FSHD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Restem, LLC. (Industry)
Collaborators: Solve FSHD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RES001-FSHD-01
Record Dates: First submitted 2025-07-03; First posted 2025-07-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: FSHD - Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: ULSC first; Placebo second (Experimental): Group 1 will receive a dose of 1 x 10^8 ULSC through IV administration on Day 0 and Month 3 (two doses, 2 x 10^8 ULSC in total from both doses). They will then cross-over to Placebo IV administrations on Month 6 and Month 9.
  Interventions: Biological: ULSC; Biological: Placebo
- Group 2: Placebo first; ULSC second (Experimental): Group 2 will receive Placebo IV administrations on Day 0 and Month 3. They will then cross-over to receive 1 x 10^8 ULSC IV administrations on Month 6 and Month 9 (2 x 10^8 ULSC in total).
  Interventions: Biological: ULSC; Biological: Placebo

INTERVENTIONS:
Biological: ULSC — Allogeneic umbilical-cord lining stem cells (ULSC) are cryopreserved and supplied in vials to be thawed and prepared for infusion at point of use. Each dose of 1 x 10^8 ULSC will be added to into 250 sterile saline for infusion (total volume of 260 mL volume).
Biological: Placebo — The Placebo will be 250 ml of sterile saline for IV administration.

SUMMARY:
The goal of this clinical trial is to learn about how an umbilical cord lining-derived stem cell product (ULSC) performs when treating Facioscapulohumeral Muscular Dystrophy (FSHD) 1 or 2. It will assess safety and preliminary efficacy in relieving symptoms of FSHD with ULSC administered in two intravenous (IV) doses of 100 million cells per dose.

The main questions that this study plans to answer are:

* Is ULSC as safe as placebo (a look-alike saline without cells) in repeated IV infusion?
* Does ULSC improve symptoms of FSHD after each dose? Researchers will compare ULSC to placebo.

Participants will:

* Have been diagnosed with FSHD of a Ricci clinical severity score 3 or more.
* Participate in this study for total duration of 21 months with 11 in-person visits and 5 virtual visits.
* Visit the clinic for a total of 4 IV infusions (250 mL) 3 months apart.
* Receive 2 doses of ULSC and 2 doses placebo in either of two sequences, as assigned: ULSC first (Day 0 and Month 3) and placebo second (Month 6 and Month 9), or placebo first (Day 0 and Month 3) and ULSC second (Month 6 and Month 9).
* Return for follow-up visits after each dose and up to 12 months after final dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥15 years old.
* Diagnosis of genetically confirmed FHSD 1 or FSHD 2.
* Participants should have a Ricci clinical severity score of ≥3 (range is out of 0-10), at screening, and must be independently ambulatory at the time of the study.
* Participant will have the ability to comply with the requirements of the study, including MRI.
* All participants of reproductive age/capacity will be required to use adequate contraception, defined as two forms of highly effective contraceptives, with any partners during the study period and for at least three months beyond the study period for safety.
* Participant will have the ability to understand and provide written informed consent.
* For those participants who are on drug(s) or supplements that may affect muscle function, as determined by the Investigator, participants must be on a stable dose of that drug(s) or supplement for at least 3 months prior to the first dose of study drug and remain on that stable dose for the duration of the study. This includes the following drug category:

  o Immunomodulatory agents, including targeted biological therapies.
* Reduced upper arm strength as measured by the Performance of Upper Limb score of ≤5.
* Current and up-to-date immunizations.
* Total relative reachable surface area (RSA) (Q1-Q4) without weight in the dominant upper extremity assessed by reachable workspace (RWS) ≥ 0.2 and ≤ 0.7.
* No contraindications to MRI.
* Hematocrit of ≤ 50%
* Prostate-specific antigen ≤ 4.0 ng/mL (or ≤ 3.0 ng/mL if the participant has a first-degree relative with prostate cancer)
* Fasting blood glucose <126 mg/dL

Exclusion Criteria:

* Hypersensitivity to study product components including history of hypersensitivity to dimethyl sulfoxide (DMSO).
* Active cancer or prior diagnosis of cancer within the past year (patients with basal and squamous cell cancer of skin will not be excluded).
* Any other condition that, in the judgment of the Investigator or Sponsor, would be a contraindication to enrollment, study product administration, or follow-up.
* Treatment with an investigational product within three months prior to randomization.
* Known active opportunistic or life-threatening infections including Human Immunodeficiency virus (HIV) and hepatitis B or C.
* Known active or inactive tuberculosis infection.
* Use of a product that putatively enhances muscle growth or activity on a chronic basis within 4 weeks before baseline
* Orally administered cytochrome P450 (CYP3A4) substrates and multidrug and toxin extrusion (MATE) and organic anion transporter (OAT)3 substrates are not permitted as concomitant therapy.
* Statin treatment initiation or significant adjustment to statin regimen within 3 months before baseline (stable, chronic statin use is permissible).
* Rapamycin treatment within 3 months before baseline.
* Evidence of an alternative diagnosis other than FSHD or a coexisting myopathy or dystrophy, based on prior muscle biopsy or other available investigations.
* Muscle biopsy within 30 days before baseline.
* A systolic blood pressure over 160 or a diastolic pressure over 100
* Heavy alcohol use (greater than 50g/day)
* Current testosterone or HGH use
* Current use of medications that interfere with the growth hormone or gonadal endocrine axis.
* Pregnant of lactating participants.
* Concomitant severe cardiac, pulmonary disease, active infection, or other conditions that preclude assessment of safety and efficacy of the study product.
* Anticipated need for surgery during the trial period.
* A history of prevalent noncompliance with medical therapy.
* Recipient of an organ transplant.
* Neutropenia (absolute neutrophil count <1,800/mm^3 [or <1,000/mm^3 in African-American participants]).
* Severe impairment in renal function (estimated glomerular filtration rate <30 ml/kg*min).
* Recent of planned use of vaccination with live attenuated viruses.
* Condition that would impair an assessment of muscle strength, including neurological disorders such as Parkinson's disease or severe musculoskeletal condition.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) and Serious Adverse Events (SAEs) that begin during or following treatment infusion. | 7 days and 30 days after each infusion, as well as 6 months after the final dose for each period (Month 9 and Month 15).
  Cumulative listing of all AEs/SAEs with descriptive statistics for categorical variables and count variables with emphasis on All SAEs and AEs/SAEs suspected to be treatment infusion-related.

SECONDARY OUTCOMES:
Facioscapulohumeral Muscular Dystrophy Composite Outcome Measure (FSHD-COM) | Baseline, 7, and 30 days after each infusion, as well as 6 months after the final dose for each period (Month 9 and Month 15).
  FSHD-COM score, which is based on objective markers of disease activity, will be assessed. The FSHD-COM is an 18-item physician-administered instrument. The body regions represented are leg function, shoulder and arm function, trunk function, hand function, and balance/mobility. Each component is scored on a 0-4 scale (0 = normal) out of a possible 72 points.
Muscle Fat Fraction (MFF) | Baseline to Month 6 and Month 12.
  Change from baseline in Muscle Fat Fraction (MFF, %) as a measure of infiltration of fat in muscle; this is assessed by Musculoskeletal (MSK) Magnetic Resonance Imaging (MRI)
Lean Muscle Volume (LMV) | Baseline to Month 6 and Month 12.
  Change from baseline in Lean Muscle Volume (LMV, cu cm or Liter) as a measure of infiltration of fat in muscle; this is assessed by Musculoskeletal (MSK) Magnetic Resonance Imaging (MRI).
Patient-Reported Quality of Life Outcome Assessed by PROMIS-57 | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 12-month timepoints.
  Change in level of disease activity as reflected in patient-reported quality of life outcome assessed by using PROMIS-57. The PROMIS-57 is a questionnaire developed by the NIH PROMIS initiative that generates scores for physical function and the impact of physical limitations on daily life.
Patient-Reported Pain Assessed by Visual Analogue Scale (VAS 10) | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 12-month timepoints.
  Change in level of patient-reported pain using Visual Analogue Scale (VAS 10) with 0 being no pain and 10 being the worst pain.
Patient-Reported Quality of Life Outcome Assessed by Activity Limitations for Patients with Upper and/or Lower Limb Impairments (ACTIVLIM) | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 12-month timepoints.
  Change in patient-reported quality of life by using ACTIVLIM 18-item questionnaire (total score scale from 0 to 36) that assess activity limitations of daily living with higher score indicating better function.
Patient-Reported Quality of Life Outcome Assessed by 5-Level EQ-5D Version (EQ-5D-5L) | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 12-month timepoints.
  Change in patient-reported quality of life by using EQ-5D-5L, which is a standardized measure of health status developed by the EuroQol Group in order to provide a measure of health that is converted to a single index value.
Patient-Reported Disease Activity & Quality of Life Outcomes Assessed by Domain Delta | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 12-month timepoints.
  Change in level of disease activity as reflected by patient-reported disease and quality of life outcomes by using Domain Delta 14-item questionnaire, which uses a 5-point scale ranging from much worse to much better. The Domain Delta is an instrument developed to assess quality of life and how disease has changed since last visit.
Patient-Reported Disease Activity & Quality of Life Outcomes Assessed by Upper Extremity Functional Index 15 (UEFI) | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 12-month timepoints.
  Change in level of disease activity as reflected by patient-reported disease and quality of life outcomes by using UEFI. The UEFI is a validated patient reported measure for adults with upper extremity dysfunction. UEFI is 20-item questionnaire with 5 possible answers ranging from 0 to 4 and a maximal score of 80. Higher scores indicate better function.
Patient-Reported Disease Activity & Quality of Life Outcomes Assessed by Facial Disability Index (FDI) for physical facial function | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 12-month timepoints.
  Change in level of disease activity as reflected by patient-reported disease and quality of life outcomes by using FDI. The FDI physical score is a short 5 item questionnaire which assesses the physical impact of facial weakness. The answers are converted to a score (scale of 0 to 100) with a higher score indicating better function.

OTHER OUTCOMES:
Iowa Oral Performance Instrument (IOPI) Scores | At each clinical visit from baseline and up to Month 12.
  Change from baseline in IOPIs at each clinical visit. Researchers have used this device in many studies to measure oral strength (kPa) with excellent inter-rater reliability.
Cardiopulmonary Exercise Testing (CPET) Assessment | From baseline to Month 6 and Month 12.
  Change from baseline in the Rating of Perceived Exertion (RPE, Borg Scale) assessed in CPET at each clinical visit.
Tissue Oxygenation Assessed by Near-Infrared Spectroscopy (NIRS) during Cardiopulmonary Exercise Testing (CPET) | From baseline to Month 6 and Month 12.
  Change from baseline of tissue oxygenation during CPET with noninvasive and continuous monitoring of regional tissue oxygenation (rSO2) using NIRS at each clinical visit.
FSHD-COM Subscales | At each clinical visit from baseline and up to Month 15.
  Change from baseline for FSHD-COM subscales assessed at each clinical visit.
Inflammatory and Immune Markers | Between baseline and the 6-month timepoint (prior to third administration), and between the 6-month and 15-month timepoints.
  Changes in the levels of inflammatory and immune biomarkers measured in plasma samples using Luminex based assays (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: John W Day, MD, PhD, Principal Investigator — Stanford University, School of Medicine, Neuromuscular Research Division
Locations (1):
- Stanford Neuroscience Health Center, Palo Alto, California, United States